CLINICAL TRIAL: NCT00051870
Title: Role of the Prefrontal Cortex in Successful Memory Encoding
Brief Title: Brain Encoding for Memory
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030081; 03-N-0081
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Healthy
Keywords: Verbal Memory; Inhibition; Transcranial Magnetic Stimulation; Cortical Excitability; Nonverbal Memory
MeSH Terms: conditions — Inhibition, Psychological

INTERVENTIONS:
Device: Magstim Rapid Magnetic Stimulator

SUMMARY:
This two-part study will use transcranial magnetic stimulation, or TMS (see below), to explore how the brain forms memories. People remember only some of the events they experience every day, such as faces they perceive, words they read, speech they hear and interpret, and so forth. The events remembered are those that have been saved or formed in the brain. Part 1 of this study involves testing materials for Part 2, the TMS experiment. Part 2 uses TMS to examine what parts of the brain are involved in forming memories. Information gained from this study may be used in developing methods of enhancing memory in both healthy people and in patients with memory impairments.

Healthy right-handed volunteers between 18 and 35 years of age may be eligible for this study. Candidates may be screened with a medical interview and physical examination and a brief test of short- and long-term visual and verbal memory. Eligible volunteers may participate in Part 1 or Part 2 of the study, as follows:

Part 1 - Preparation of Words and Picture Materials

Participants look at several words or shapes that appear in random order on a computer screen and try to remember them as well as possible for a memory test that will be given 20 minutes later. Each image appears on the screen for 3/4 of a second, with 1-1/4-second intervals between them. For the test, words and shapes are again shown on the computer screen at the same timing and intervals. When the items appear, the subject presses one of three buttons as quickly as possible, determining if he or she has recognized the items with a high or low level of confidence. The entire procedure lasts up to 1 hour, with breaks in between. The purpose of this experiment is to find appropriate words and pictures to use as stimuli in the TMS study described below.

Part 2 - TMS Experiment

For TMS, the subject sits in a comfortable chair. An insulated wire coil is placed on the scalp, and brief electrical currents are passed through the coil, creating magnetic pulses that stimulate the brain. The pulses may cause a pulling sensation on the skin under the coil and twitching in muscles of the arm or leg. Electrodes are taped to the skin over some muscles of the hands to record the electrical activity of the muscles. Pulses are delivered in trains or short bursts of impulses, each lasting half a second. Participants receive 90 trains for a total of 900 pulses. TMS is applied during the first part of the memory study, when the words and shapes are first presented on the computer screen, but not during the second presentation for memory testing. The entire procedure takes up to 2 hours, with breaks in between.

Before the TMS session, participants undergo magnetic resonance imaging (MRI) to determine where to place the coil for TMS. For MRI, the subject lies still for up to 30 minutes at a time on a table that slides into the scanner, a narrow metal cylinder surrounded by a strong magnetic field. Earplugs are worn to muffle loud knocking sounds that occur while the scanner takes pictures. Subjects can communicate with the MRI staff at all times and can ask to stop the procedure at any time.

DETAILED DESCRIPTION:
Recent functional imaging studies showed that memory retrieval is associated with activation in the prefrontal cortex during the encoding process. However, a cause-effect link between prefrontal activity and encoding has not been demonstrated. The purpose of this protocol is to test the hypothesis that inhibitory repetitive transcranial magnetic stimulation (rTMS) over left prefrontal cortex interferes with encoding of verbal items (words) into episodic memory, thereby identifying this region as a substrate mediating verbal encoding. Identification of the role of the prefrontal cortex in verbal memory encoding is the first step to try to develop strategies to enhance such encoding processes in patients with memory impairments, an issue of relevance in neurorehabilitation.

We plan to apply rTMS over left prefrontal cortex and over two control sites, during encoding of verbal and nonverbal items into episodic memory. Normal, healthy volunteers will be studied. The outcome measure will be performance on a subsequent memory test for words presented during left prefrontal rTMS, as compared to performance for words presented during rTMS over the control sites or without rTMS. This measure will indicate if left prefrontal stimulation can disrupt memory encoding of words relative to other stimulation sites or to no stimulation.

A secondary outcome measure will be performance on a subsequent memory test for words presented during left prefrontal rTMS, as compared to performance for pictures presented during left prefrontal rTMS. This measure will indicate if disruption of left prefrontal function with TMS affects verbal and more than non-verbal memory encoding.

ELIGIBILITY:
INCLUSION CRITERIA:

INCLUSION CRITERIA:

Healthy right handed volunteers, aged 18-35 years, will be included in this protocol.

EXCLUSION CRITERIA:

Exclusion criteria for this study will be any current medical or surgical condition or psychiatric or neurological illness. Furthermore, any individual who is on medication with potential influence on nervous system function, who has a history of surgery with metallic implants or known history of metallic particles in the eye, cardiac pacemaker, neural stimulators, cochlear implants, pregnancy, or history of drug abuse, will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Squire LR, Knowlton B, Musen G. The structure and organization of memory. Annu Rev Psychol. 1993;44:453-95. doi: 10.1146/annurev.ps.44.020193.002321. No abstract available. PMID 8434894
- [Background] Tulving E, Markowitsch HJ, Craik FE, Habib R, Houle S. Novelty and familiarity activations in PET studies of memory encoding and retrieval. Cereb Cortex. 1996 Jan-Feb;6(1):71-9. doi: 10.1093/cercor/6.1.71. PMID 8670640
- [Background] Kapur S, Tulving E, Cabeza R, McIntosh AR, Houle S, Craik FI. The neural correlates of intentional learning of verbal materials: a PET study in humans. Brain Res Cogn Brain Res. 1996 Nov;4(4):243-9. doi: 10.1016/s0926-6410(96)00058-4. PMID 8957565